CLINICAL TRIAL: NCT02947386
Title: A Phase I/II Open-Label Study of Nimotuzumab in Combination With Nivolumab in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Nimotuzumab and Nivolumab in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 281616; NCI-2016-01476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 281616 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: EGFR Gene Mutation; Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nimotuzumab; TheraCIM; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, nimotuzumab) (Experimental): Patients receive nivolumab IV over 60 minutes and nimotuzumab IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nimotuzumab; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nimotuzumab — Given IV
  Other Names: Thera-CIM-hr3; TheraCim hR3; Theraloc
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase I/II trial studies the best dose and side effects of nimotuzumab when giving together with nivolumab and to see how well they work in treating patients with non-small cell lung cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Monoclonal antibodies, such as nimotuzumab and nivolumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicities (DLT) and estimate the maximum tolerated dose (MTD) of nimotuzumab combined with nivolumab in the therapy of advanced non-small cell lung cancer (NSCLC) in order to establish the recommended phase II dose (RP2D). (Phase I)

II. To evaluate the 12 month overall survival of nimotuzumab in combination with nivolumab in patients with advanced NSCLC. (Phase II)

SECONDARY OBJECTIVES:

I. Examine the safety and tolerability profile of nivolumab in combination with nimotuzumab in NCSLC . (Phase I)

II. To evaluate the safety and the tolerability of nimotuzumab in combination with nivolumab using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0). (Phase I)

III. Determine the immune analysis profile of nivolumab in combination with nimotuzumab. (Phase I)

IV. Examine the efficacy of the study combination utilizing irRECIST guidelines. (Phase I)

V. Overall response rate (ORR) per the immune-related Response Evaluation Criteria in Solid Tumors irRECIST. (Phase I)

VI. Progression-free survival (PFS) rate at 1 year. (Phase I)

VII. Progression-free survival (PFS). (Phase I)

VIII. Overall survival (OS). (Phase I)

IX. Disease control rate (DCR) and stable disease (SD). (Phase I)

X. To evaluate the safety profile of Nimotuzaumab in combination with Nivolumab in NCSLC using the CTCAE V. 4.

XI.To evaluate the efficacy of nimotuzumab in combination with nivolumab in patients with advanced NSCLC compared to historic outcomes of nivolumab alone, as determined by secondary measures of efficacy, including: overall response rate (ORR) per irRECIST. (Phase II)

XII. To evaluate the efficacy of nimotuzumab in combination with nivolumab in patients with advanced NSCLC compared to historic outcomes of nivolumab alone, as determined by secondary measures of efficacy, including: progression-free survival (PFS) rate at 1 year. (Phase II)

XIII. To evaluate the efficacy of nimotuzumab in combination with nivolumab in patients with advanced NSCLC compared to historic outcomes of nivolumab alone, as determined by secondary measures of efficacy, including: progression-free survival (PFS). (Phase II)

XIV. To evaluate the efficacy of nimotuzumab in combination with nivolumab in patients with advanced NSCLC compared to historic outcomes of nivolumab alone, as determined by secondary measures of efficacy, including: overall survival (OS). (Phase II)

XV. To evaluate the efficacy of nimotuzumab in combination with nivolumab in patients with advanced NSCLC compared to historic outcomes of nivolumab alone, as determined by secondary measures of efficacy, including: disease control rate (DCR) and stable disease (SD). (Phase II)

TERTIARY OBJECTIVES:

I. Examine the relationship of EGFR expression in tissue to PFS, OS, ORR and adverse events (AE). (Phase I)

II. Examine the relationship of infiltrating CD4+ and CD8+ T cells and other immune and genetic markers, and their associated PD-1, CD45RA or CD45RO levels; PD-L1 expression within both neoplastic and non-neoplastic stromal elements of the tumor microenvironment to PFS, OS, ORR and AE. (Phase I)

III. Comparison of response assessment criteria for a prospective analysis; irRECIST response assessment; irRC. (Phase I)

IV. Examine the relationship of EGFR expression in tissue to PFS, OS, ORR and AE. (Phase II)

V. Examine the relationship of infiltrating CD4+ and CD8+ T cells and other immune and genetic markers, and their associated PD-1, CD45RA or CD45RO levels. (Phase II)

VI. Examine the relationship of PD-L1 expression within both neoplastic and non-neoplastic stromal elements of the tumor microenvironment to PFS, OS, ORR and AE. (Phase II)

VII. Comparison of response assessment criteria for a prospective analysis; irRECIST response assessment; irRC. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of nimotuzumab followed by a phase II study.

Patients receive nivolumab intravenously (IV) over 60 minutes and nimotuzumab IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients with pathologically confirmed non-small cell lung cancer
* Patients must have had progressive NSCLC after first-line platinum-based chemotherapy for advanced disease
* Have at least 3 months life expectancy
* Have measurable disease per RECIST 1.1 criteria present
* Patients with adenocarcinoma known to have anaplastic lymphoma kinase (ALK) rearrangements and/or epidermal growth factor receptor (EGFR) mutations that have had prior EGFR or ALK tyrosine kinase inhibitor therapy and have progressed, will also be eligible, regardless of line of therapy
* Phase I optional archival tissue/phase II mandatory archival tissue: able to provide enough biopsy tissue samples including primary diagnostic biopsy (archival), re-biopsy tissues (archival from time of disease progression/recurrence following first-line treatment failure) at disease progression to determine PD-L1 and EGFR expression and other biomarkers
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 x institution upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 1.5 x ULN or =< 5 x ULN if liver metastases are present
* Total serum bilirubin =< ULN; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's syndrome
* Troponin-I, CK-MB +< BNP <200pg/ml
* LVEF >= LLN
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Active autoimmune disease that has required systemic treatment in past 2 years; use of inhaled corticosteroids is allowed
* Phase II only: history of other malignancies are allowed as long as the current disease stage that did not require active treatment with concomitant systemic cytotoxic chemotherapy, targeted therapy, investigational or biologic therapy (e.g., anti-CTLA4 or HER2 monoclonal antibodies) within 12 months prior to study registration and, is not likely to require systemic therapy in the next 12 months; hormone-related therapies (e.g., somatostatin analogues, etc.) are allowed on a case-to-case basis upon discussion with principal investigator
* Active clinically serious infections requiring antibiotics, antiviral or antifungal agents
* Symptomatic brain metastases; uncontrolled pleural effusion, seroperitoneum, or pericardial effusion
* Has had any major surgery, chemotherapy, or radiotherapy within the previous 4 weeks; gamma knife radiosurgery for brain metastases within less than 2 weeks
* Receiving other anti-cancer medical treatment during the study outside of the nimotuzumab or nivolumab
* Clinically significant interstitial pulmonary disease or known diagnosis of interstitial lung disease (ILD)
* Has known immunosuppressive disease (e.g. human immunodeficiency virus [HIV], acquired immune deficiency syndrome [AIDS])
* Patient has known hypersensitivity to the components of the study drugs or their analogs
* Patient with uncontrolled cardiac disease or cardiac dysfunction, including any of the following:

  * History of uncontrolled angina pectoris that does not respond to medical intervention
  * Symptomatic pericarditis or myocardial infarction within 12 months prior to study entry that did not respond to treatment
  * History of documented congestive heart failure (New York Heart Association functional classification III or IV)
  * Documented cardiomyopathy
  * Uncontrolled hypertension defined by: systolic blood pressure (SBP) >= 160 mmHg and/or diastolic blood pressure (DBP) >= 100 mmHg
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
DLT as graded by NCI CTCAE version 4.0 (Phase I) | Up to 28 days
  No formal analyses of DLTs are planned. Participants who do not have a DLT and who do not complete a full cycle of treatment will be considered non-evaluable for DLT.
ORR defined as complete response (CR) + partial response (PR) divided by number of patients as assessed by RECIST version 1.1 (Phase II) | Up to 3 years
  Will be calculated as the number of patients with a confirmed complete or partial response divided by the total number of patients. The 95% confidence interval for ORR (CR + PR) will be presented based on the Wilson Score method as irRC response.

SECONDARY OUTCOMES:
Incidence of adverse events assessed by NCI CTCAE version 4.0 (Phase I and II) | Up to 30 days after the last dose of study treatment
  The frequency of AEs will be tabulated by grade across all dose levels and cycles. All patients who receive any study treatment will be considered evaluable for toxicity.

OTHER OUTCOMES:
EGFR expression in tumor tissue (Phase I and II) | Up to 3 years
  Examined using Kaplan-Meier plots and log-rank tests or proportional hazards models for time-to-event data, and presentation of frequencies and proportions and exact tests for binary and categorical data.
PD-L1 expression in tumor tissue (Phase I and II) | Up to 3 years
  Examined using Kaplan-Meier plots and log-rank tests or proportional hazards models for time-to-event data, and presentation of frequencies and proportions and exact tests for binary and categorical data.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Dy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States